CLINICAL TRIAL: NCT06102434
Title: Safety Profile of 25 mg Psilocybin in Individuals With Cocaine Use Disorder
Brief Title: Safety Profile of Psilocybin for Cocaine Use Disorder
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Conor Murray, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-002081
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 25 mg psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Five oral capsules containing 5 mg of psilocybin each

SUMMARY:
The purpose of this study is to establish the safe administration of psilocybin in individuals with cocaine use disorder in terms of cardiovascular (e.g., heart rate) and subjective (e.g., mood) effects. The study's subject population consists of men and women between the ages of 21 and 55 from the Los Angeles area that meet criteria for cocaine use disorder and express an interest in ceasing cocaine use. 25 mg oral psilocybin will be administered to 10 individuals (separately) during a single laboratory visit. The laboratory visit will take place from 9 am until 3 pm within a comfortable, living room like environment. Within this study session room, participants will be accompanied by two clinicians. Participants will then consume the psilocybin capsule, and thereafter will be encouraged to lie down on a couch and introspect on the experience. At one-hour intervals following ingestion, participants will be tested briefly for changes in heart rate, blood pressure, and subjective effects. No blood draws, behavioral assessments, or neuroimaging is included in the study. Following the laboratory visit, investigators will check-in on participants remotely, after 48 hours, and 10, 50, and 90 days from the psilocybin session.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index from 18.5 - 34kg/m^2
* Score of at least 3 on the Severity of Dependence Scale
* Desire to cease cocaine use as indicated by a goal of complete cocaine abstinence on the Thoughts about Abstinence Questionnaire
* At least 1, but not more than 10 total lifetime use of a classical psychedelic (5-HT2a agonist)
* 0 use of a classical psychedelic in the last year

Exclusion Criteria:

* History of serious adverse events in response to classical psychedelics including history of Hallucinogen Persisting Perceptive Disorder
* Abnormal electrocardiogram based on testing at study entrance
* A resting heart rate greater than 90 bpm
* Current hypertension (exceeding 140 systolic and 90 diastolic at resting)
* Current use of antidepressants or other serotonergic-affecting substances
* History of cardiac conditions
* History of hepatic or renal impairments
* History of stroke or Transient Ischemic Attack
* Epilepsy or history of seizures
* Immediate family or personal history of psychosis, bipolar disorder, or schizophrenia
* Anxiety or mood disorders determined by the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-V)
* Must not meet DSM-V criteria for any substance use disorders other than cocaine, caffeine, or nicotine
* Must not meet DSM-V criteria for borderline personality or dissociative disorders
* Current suicidal ideation or lifetime history of suicide attempts
* Arrest for a violent offense
* Any clinical condition, history of illness, or laboratory results that may place participants at greater risk as judged by the study physician
* Women will not be eligible if trying to get pregnant, pregnant, or lactating

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart rate | From pre-dose through one-hour intervals post-dose until heart rate has returned to within 20% of the pre-dose measure, or after a minimum of 6 hours.
  Beats per minute measured with blood pressure monitor.
Blood pressure | From pre-dose through one-hour intervals post-dose until blood pressure has returned to within 20% of the pre-dose measure, or after a minimum of 6 hours
  Systolic and diastolic blood pressure measured with blood pressure monitor.
Self-reported drug effects | From pre-dose through one-hour intervals post-dose over a 6-bour period.
  Average and peak subjective ratings of drug effects associated with mood measured using visual analogue scales (VAS; 1-100 mm).

SECONDARY OUTCOMES:
Self-reported cocaine craving | 48 hours and 10, 50, and 90 days after psilocybin administration.
  Average subjective ratings of cocaine craving measured using Cocaine Craving Questionnaire-Brief. Each item on the 10 item questionnaire is scored on a scale ranging from 1 for "Strongly Disagree" to 7 for "Strongly Agree," with higher scores indicating greater cocaine craving.
Self-reported mood ratings | 48 hours and 10, 50, and 90 days after psilocybin administration.
  Average subjective ratings of Depression, Anxiety, Stress measured using Depression, Anxiety and Stress scales of the Depression Anxiety Stress Scale (DASS-21). Each scale consists of 7 items rated from 0 to 3, with higher scores indicating greater Depression, Anxiety, or Stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided